CLINICAL TRIAL: NCT00723684
Title: ADHD and EEG-neurofeedback. A Single-blind Randomized Placebo-controlled Treatment Study.
Brief Title: Project Attention Deficit Hyperactivity Disorder (ADHD) and Electroencephalography (EEG)-Neurofeedback THERapy
Acronym: PANther
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Prof. Jan Buitelaar, professor dr., Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NF1
Record Dates: First submitted 2008-07-28; First posted 2008-07-29 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-03

CONDITIONS: ADHD
Keywords: ADHD; Children; EEG-Neurofeedback
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo group (Placebo Comparator): This group will receive no real EEG-Neurofeedback.
  Interventions: Other: Placebo EEG Neurofeedback
- NF group (Experimental): This group will receive real EEG-Neurofeedback
  Interventions: Other: EEG-Neurofeedback

INTERVENTIONS:
Other: Placebo EEG Neurofeedback — The placebo EEG-neurofeedback group will get an identical procedure as the real EEG-Neurofeedback, but with feedback on a EEG signal simulation. The placebo group will not be rewarded on their real-time EEG but on a random, simulated EEG; known to be effective for this purpose (Utrecht University, study in progress).
  In the protocol selection the electrode position and rewarding versus inhibition of the treatment frequency band or bands will be individually created. The first 30 seconds of the treatment will start on a predetermined fixed threshold value for all treatment subjects.
  Arms: Placebo group
Other: EEG-Neurofeedback — The EEG-neurofeedback group will receive feedback on their real-time EEG-signal (brain activity). The treatment group will be rewarded, by brightening (i.e. not being blackened of) the feedback screen. Rewards will be given to the subjects when their digitally filtered frequency EEG activity meets the criteria in the 'percentage time over threshold' parameter. The 'percentage time over threshold' parameter will be auto-adjusted on the digitally filtered real-time EEG every 30 seconds, and the percentage parameter will be kept as a constant over all participants during the entire study (i.e. not adjusted during treatment based on individual capabilities).
  Arms: NF group

SUMMARY:
Background:

Electroencephalography (EEG)-neurofeedback has been shown to offer therapeutic benefits to patients with ADHD in several mostly uncontrolled studies with relatively small sample sizes. It is unknown how EEG-neurofeedback affects brain functioning and exerts therapeutic effects in ADHD. This study is designed to examine the efficacy and safety of EEG-neurofeedback in a scientific rigorously way and to study the underlying neurobiological mechanisms of EEG-neurofeedback.

Objectives:

1. To investigate the efficacy of EEG-neurofeedback in reducing behavioral symptoms of ADHD.
2. To investigate whether EEG-neurofeedback is able to improve neurocognitive functioning.
3. To investigate whether EEG-neurofeedback is able to improve neural functioning.

Study design:

Double-blind randomized placebo-controlled treatment study.Study population: 120 subjects with ADHD (age 8-15, IQ of 80 or more). Intervention: 60 subjects with ADHD receive 30 sessions EEG-neurofeedback, and 60 subjects with ADHD receive placebo EEG-neurofeedback.

Main study parameter: ADHD-DSM-IV rating scale, rated by the investigator.

Hypothesis:

The hypothesis is EEG-Neurofeedback can reduce symptoms of ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis ADHD, classified by the (Diagnostic and Statistical Manual of Mental Disorders, 2000)
* Age between 8 and 15
* A full scale IQ of more than 80
* Psychopharmaca- naïve or -free, or using a stable dosage of psychostimulants or atomoxetine but still with room for improvement (defined by an average score of more than 1 on ADHD-DSM-IV rating scale).
* Deviant EEG of more than 1.5 standard deviation compared to the database

Exclusion criteria:

* Currently intensive (i.e. weekly) individual or group psychotherapy
* Regular use of medication other than psychostimulants or atomoxetine
* Diagnosis of one or more of the following comorbid psychiatric disorders:
* Major depression
* Bipolar disorder
* Psychotic disorder
* Chronically motor tic disorder or Gilles de la Tourette
* Conduct disorder
* Autism spectrum disorders
* Eating disorders
* Neurological disorders (e.g. epilepsy) currently or in the past
* Cardiovascular disease currently or in the past
* Participation in another clinical trial simultaneously
* EEG-neurofeedback training in the past
* Use of alcohol or drugs

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2008-07; Primary Completion 2012-07 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
ADHD criteria according to the DSM-IV-TR rated by the investigator. | before, after 10, 20, 30 sessions and after half a year

SECONDARY OUTCOMES:
side-effects by Score on the adapted Pittsburgh side effects rating scale | before, after 10, 20, 30 sessions

CONTACTS AND LOCATIONS:
Overall Officials: J.K. Buitelaar, Professor, Principal Investigator — UMC St. Radboud and Karakter
Locations (2):
- Netherlands (2):
  - FC Donders Centre for Cognitive Neuroimaging, Nijmegen, Gelderland
  - Karakter Nijmegen, Nijmegen, Gelderland

REFERENCES:
- [Derived] Vollebregt MA, van Dongen-Boomsma M, Buitelaar JK, Slaats-Willemse D. Does EEG-neurofeedback improve neurocognitive functioning in children with attention-deficit/hyperactivity disorder? A systematic review and a double-blind placebo-controlled study. J Child Psychol Psychiatry. 2014 May;55(5):460-72. doi: 10.1111/jcpp.12143. Epub 2013 Oct 30. PMID 24168522
- [Derived] van Dongen-Boomsma M, Vollebregt MA, Slaats-Willemse D, Buitelaar JK. A randomized placebo-controlled trial of electroencephalographic (EEG) neurofeedback in children with attention-deficit/hyperactivity disorder. J Clin Psychiatry. 2013 Aug;74(8):821-7. doi: 10.4088/JCP.12m08321. PMID 24021501